CLINICAL TRIAL: NCT04917614
Title: Effect of Transcutaneous Electrical Acupoint Stimulation on Obstetric Quality of Recovery-10 After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TEAS and ObsQoR-10
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Recovery
Keywords: ObsQoR-10T; recovery; ceserean; postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group teas (Active Comparator): Patients in the TEAS group will receive preoperative TEAS for 30 min before the spinal anesthesia at Hegu (LI4), Neiguan (PC6), and Zusanli (St 36) with an electronic acupuncture device.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation
- Control Group (Sham Comparator): In the sham group, the patients were connected to the electronic acupuncture, but electronic stimulation was not applied.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Acupoint Stimulation — Transcutaneous Electrical Acupoint Stimulation

SUMMARY:
The primary aim of this prospective and randomized trial is to investigate the effect of TEAS on postoperative recovery using the Obstetric Quality of Recovery-10 questionnaire in patients undergoing elective cesarean section.

DETAILED DESCRIPTION:
Acupoint stimulation is postulated to modulate neurological signal transmission through afferent nociceptive pathways. Acupoint stimulation has been associated with positive effects on perioperative symptoms such as nausea, pain, and sleep disturbance. Transcutaneous electrical acupuncture point stimulation (TEAS) is an acupuncture treatment developed by combining traditional Chinese acupuncture with transcutaneous electrical nerve stimulation. TEAS has proven to be effective in postoperative pain and nausea-vomiting by applying a current of different frequencies, intensities, and waveforms through electrodes adhering to the skin. Using TEAS may relieve perioperative symptoms without increasing the risk of drug-related adverse events and alleviate and improve the patient's health condition, including the postoperative perspective.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean operation
* Able to give informed consent

Exclusion Criteria:

* Patients with neurological or psychological diseases
* patients with chronic analgesic and antidepressant drug use
* Patients unable to communicate
* Patients previously treated with TEAS or acupuncture,
* Patients with heart failure and have pace-maker,
* patient with local infection in the TEAS area

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2021-07-18 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery | The first 24 hours postoperatively
  Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Betul Kozanhan, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No